CLINICAL TRIAL: NCT02786784
Title: The Role of Arthrogenic Muscular Inhibition in Patellofemoral Pain and the Response to an Exercise Programme
Acronym: PFP-Inhibit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Salford (Other)
Collaborators: Northern Care Alliance NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Henrike Greuel, PhD student, Principal Investigator, University of Salford
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRAS 194530
Record Dates: First submitted 2016-05-23; First posted 2016-06-01 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: PFP; Patellofemoral Pain; Anterior Knee Pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- healthy control (Other): patients with patellofemoral pain
  Interventions: Other: 6 week exercise treatment

INTERVENTIONS:
Other: 6 week exercise treatment — This six-week exercise programme was developed based on the current recommendations, consisting of four exercises to strengthen gluteus medius and maximus muscle, as well as the quadriceps muscle. In addition, two exercises to stretch the hamstrings muscles and to increase the ankle dorsi range of motion were included.

SUMMARY:
Patellofemoral pain (PFP) is the most diagnosed condition in individuals with knee complaints. Studies revealed that one third of individuals with PFP suffer from persistent complaints, indicating that current treatments fail to prevent the chronicity of symptoms. Considering that current treatment-strategies of patients with PFP seem to be unable to avoid the development of chronic symptoms, the question arises if the underlying factors of PFP are understood sufficiently. Current research focuses predominantly on muscle strength assessment by means of a maximum voluntary contraction (MVC), even though, weakness might not only be caused by a reduced voluntary contraction but also by an involuntary ability to contract the muscle fully, which is named arthrogenous muscular inhibition (AMI). Although AMI has been proven to be present in a wide range of knee joint pathologies to date it remains unclear whether patients with PFP are weak or inhibited. It remains also unclear if there exists a causal link between AMI and biomechanical alterations.

Previous studies investigated the influence of exercise treatment on muscular strength, function and pain. However, to date no study investigated the influence of the currently recommended exercise treatment on AMI. Thus, the analysis of the effect of a 6 week exercise treatment might yield further insights if a specific exercise treatment can reduce AMI, improve functional performance and reduce pain.

Methods: The investigators will invite 40 participants with PFP and 40 healthy controls to take part in the study. As a basis investigation kinematic, kinetic measures, and surface electromyographic (sEMG) of 4 lower limb muscles will be taken during functional tasks. Muscle strength and AMI of the quadriceps, muscle flexibility, and a posture assessment of the patella as well as the foot will be carried out. All participants with PFP will then receive a 6 week exercise programme to follow. After six weeks, the participants with PFP will attend the Salford university, where they will be reassessed.

Expected outcomes: The study will investigate if AMI is present in participants with PFP and if AMI is directly linked to functional performance. In addition this study will investigate if a specific exercise treatment can reduce AMI and improve functional performance.

DETAILED DESCRIPTION:
Procedures The testing will be performed in the human performance laboratory at the University of Salford, Manchester. Upon arrival at the laboratory, the participants will be briefed through the study and the objectives of the investigations and the study equipment will be explained to them. They will be asked to sign the informed consent form, a health history questionnaire. The health history questionnaire consists of 13 questions investigating potential risks associated with the study.

The individual will then be asked to change into their shorts and a comfortable t-shirt.

Strength and arthrogenic muscle inhibition:

The muscular inhibition of the quadriceps will be assessed, during a maximal isometric contraction (MVIC) of the quadriceps with the interpolated twitch technique. The participants will perform 5 times a maximal contraction of their knee extensor and additional electrical stimulation will be applied, which will be performed on an isokinetic dynamometer (Kin-Com) with a knee flexion angle of 90°. Then the participant will be asked to perform 5 times an eccentric quadriceps contraction at the angular velocity of 60 degrees/ second, through the full available range of motion (ROM) from 90 degrees knee flexion to maximum knee extension, while the quadriceps torque will be measured.

Questionnaires:

The participants with PFP will then be asked to fill in 3 different questionnaires:

the KOOS, the AKPS/ Kujala score, and the Tampa Scale of Kinesiophobia.

After this recovery break, the posture and flexibility investigation will be executed. The examination of the foot posture will be performed by using the 6-item foot posture index (FPI-6). The patella alignment includes a lateral - medial displacement/ lateral -medial tilt), and a lateral-medial displacement assessment.

Flexibility:

The flexibility of the hamstrings and the soleus muscle will be assessed.

Biomechanics:

Following this, the researcher will attach 40 retro-reflective markers to the skin of the lower limb on both legs and attach surface electromyographic electrodes to four muscles as in figure 4 on both legs. The electrode placement will be performed according to the SENIAM guidelines. Suface EMG (sEMG) data will be collected of vastus medialis, vastus lateralis, biceps femoris and semitendinosus will be synchronised with the motion capture system on Qualisys.

After a static 3-dimensional image from ten infra-red cameras will be obtained. The 3D kinematics of the ankle, knee, and hip joint and ground reaction forces (GRF) will be recorded for each participant during a running, a single leg squat and a step down task.

Treatment:

The 6 week treatment will be exclusively conducted by physiotherapists at the Salford Royal Hospital (Salford Royal NHS Foundation Trust, SRFT).

Physiotherapist from the Salford Royal hospital will introduce the treatment programme to the participants. Additionally, each participants will receive a booklet with a detailed description of the treatment programme, as well as access to a password protected website (VIMEO) to watch the videos of all exercises.

Assessment of the treatment outcomes after 6 weeks At the end of the 6 weeks exercise intervention, the participants with PFP will then attend the human performance laboratory at the University of Salford. The muscle strength, AMI, flexibility, posture assessment, as well as the clinical assessment of running and a step down task of each individual will be measured to investigate the change in AMI and functional performance due to the treatment.

ELIGIBILITY:
Inclusion Criteria for patients with PFP:

1. Reproducible pain with at least two of these activities: ascending or descending stairs or ramps, squatting, kneeling, prolonged sitting, hopping/ jumping, isometric quadriceps contraction or running
2. Clearly defined pain location in the peripatellar region
3. Reports of pain greater than 1 month duration.
4. They are able to perform squatting, running and MVC task- Participant response
5. Age range: 18-45 years old

Inclusion criteria for healthy volunteers:

1. Healthy and without any previous lower limb injuries
2. The participant is able to perform squatting, running and MVC task

Exclusion Criteria for all participants:

1. Previous history of knee surgery
2. Previous history of (traumatic) patella dislocation or instability
3. Previous history of ligamentous instabilities
4. Previous history of traumatic, inflammatory or infectious pathology in the lower extremity
5. Previous history of internal derangement or other causes
6. Previous diagnosed degenerative conditions in the knee
7. Exclusion if patients cannot perform running, step down, or MVC task.
8. Exclusion criteria for the healthy control group are: clinical evidence of other knee injury or knee pain, and current significant injury affecting other lower extremity joints.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-09 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Extent of the arthrogenic muscle inhibition (AMI) | 6 weeks
  AMI will be calculated from the ratio:
  AMI = (resting twitch size in Nm/ twitch size during MVC in Nm)*100 AMI will be expressed in %. The differences between the baseline measurements and the measurements after 6 weeks of treatments will be investigated in participants with PFP.
quadriceps/ hamstrings cocontraction | 6 weeks
  The cocontraction of the quadriceps (vastus medialis and lateralis) and the hamstring (biceps femoris and semitendinosus) was calculated by the formula developed by Heiden et al. 2009, whereby 0 expresses no cocontraction and 1 a complete cocontraction. The cocontraction will be calculated for for the early, mid, late stance phase, the single leg squat and single leg step down task. Differences between the baseline of participants with PFP and after 6 weeks after the treatment will be investigated.
  Furthermore, the correlation between the external knee adduction moment (EKAM) to AMI will be investigated.
Presence of the break phenomenon | 6 weeks
  The break phenomenon is defined as a trace dip during the eccentric quadriceps phase, which exceeds more than 10% of the pre-break moment. The break phenomenon will be defined as either: present or not present. The differences between the baseline measurements and the measurements after 6 weeks of treatments will be investigated in participants with PFP.
Maximal knee adduction angle | 6 weeks
  The maximal knee adduction angle will be given for the early, mid, late stance phase, the single leg squat and single leg step down task and will be expressed in degrees. The differences between the baseline measurements and the measurements after 6 weeks of treatments will be investigated in participants with PFP.
Maximal knee adductor moment (EKAM) | 6 weeks
  The maximal knee adductor moment will be given as % of the bodyweight (BW). The maximal EKAM will be investigated for early, mid, late stance phase, the single leg squat and single leg step down task. The differences between the baseline measurements and the measurements after 6 weeks of treatments will be investigated in participants with PFP.
the knee adduction angular impulse (KAAI) | 6 weeks
  knee adduction angular impulse is defined as the integral of the knee adduction moment-time curve. The normalised KAAI will be given as % of the bodyweight (BW). The KAAI will be given for early, mid, late stance phase, the single leg squat and single leg step down task. The differences between the baseline measurements and the measurements after 6 weeks of treatments will be investigated in participants with PFP.
Maximal knee internal rotation | 6 weeks
  The maximal knee internal rotation angle will be given for the early, mid, late stance phase, the single leg squat and single leg step down task and will be expressed in degrees. The differences between the baseline measurements and the measurements after 6 weeks of treatments will be investigated in participants with PFP.
Maximal knee internal rotation moment | 6 weeks
  The maximal knee internal rotation moment will be given as % of the bodyweight (BW). The maximal knee internal rotation moment will be investigated for early, mid, late stance phase, the single leg squat and single leg step down task and will be expressed as % of the bodyweight (BW). The differences between the baseline measurements and the measurements after 6 weeks of treatments will be investigated in participants with PFP.
Maximal hip adduction angle | 6 weeks
  The maximal hip adduction angle will be given for the early, mid, late stance phase, the single leg squat and single leg step down task and will be expressed in degrees. The differences between the baseline measurements and the measurements after 6 weeks of treatments will be investigated in participants with PFP.
Maximal hip adduction moment | 6 weeks
  The maximal hip adductor moment will be given as % of the bodyweight (BW). The maximal hip adductor moment will be investigated for early, mid, late stance phase, the single leg squat and single leg step down task and will be expressed as % of the bodyweight (BW). The differences between the baseline measurements and the measurements after 6 weeks of treatments will be investigated in participants with PFP.
Maximal hip internal rotation | 6 weeks
  The maximal hip internal rotation angle will be given for the early, mid, late stance phase, the single leg squat and single leg step down task and will be expressed in degrees. The differences between the baseline measurements and the measurements after 6 weeks of treatments will be investigated in participants with PFP.
Maximal hip internal moment | 6 weeks
  The maximal hip internal rotation moment will be given as % of the bodyweight (BW). The maximal hip internal rotation moment will be investigated for early, mid, late stance phase, the single leg squat and single leg step down task and will be expressed as % of the bodyweight (BW). The differences between the baseline measurements and the measurements after 6 weeks of treatments will be investigated in participants with PFP.

SECONDARY OUTCOMES:
temporo-spatial parameters: speed | 6 weeks
  The gait speed will be analysed and expressed as mean and SD.
temporo-spatial parameters: step length | 6 weeks
  The step length will be analysed and expressed as mean and SD.
Muscle strength: peak strength during the eccentric quadriceps task | 6 weeks
  The peak strength will be measured during the eccentric quadriceps testing (Kin Com).
Muscle strength: peak strength during the isometric quadriceps task | 6 weeks
  The peak strength will be measured during the isometric quadriceps testing (Kin Com).
KOOS, AKPS, Tampa scale questionnaires | 6 weeks
  Only patients with PFP will be asked to fill them. For each of the questionnaires a normalized score will be calculated for each subscale. The differences of the overall score will be calculated to ensure that confounding factors, such as kinesiophobia are controlled and checked.
Foot posture | 6 weeks
  The results of the 6-item foot posture index will be summarised, whereby a negative result expresses a supinated and a positive result a pronated foot.
Lateral/ medial displacement of the patella | 6 weeks
  The lateral/ medial displacement of the patella will be measured and expressed in cm.
Lateral/ medial tilt of the patella | 6 weeks
  The lateral/ medial tilt of the patella will be measured and on a scale from -2 (strongly laterally tilted) to 2 (strongly medially tilted)
Flexibility of the quadriceps | 6 weeks
  The quadriceps flexibility will be assessed by using the modified Thomas test and will be expressed in degrees of the knee flexion.
Flexibility of the hamstrings | 6 weeks
  The hamstrings flexibility will be assessed by using the active knee extension test and will be expressed in degrees of the knee flexion.
Flexibility of the ankle range of motion. | 6 weeks
  The ankle flexibility will be assessed by using the weight bearing lunge test and will be expressed in degrees of the ankle dorsalflexion and in cm, by measuring the distance of the 1st toe to the wall.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Salford, Salford, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided